CLINICAL TRIAL: NCT06950502
Title: Comparison of the Effects of Bilateral Transversus Abdominis Plane Block and Bilateral Quadratus Lumborum Block on Postoperative Analgesia in Patients Undergoing Midline Laparotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Esma Asik, Research Asistant, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAsik
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: QLB vs TAPB; Quadratus Lumborum Block; Transversus Abdominis Plane (TAP) Block
Keywords: Oblique subcostal transversus abdominis plane block; Quadratus lumborum block; Pain; Regional Anaesthesia
MeSH Terms: conditions — Bites and Stings; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus Lumborum Group (QLB) (Active Comparator): Quadratus lumborum block; after the patient was lying in the lateral decubitus position and skin asepsis of the posterior abdominal wall was provided with 10% polyvinylpyrrolidone-iodine, the ultrasound probe was moved from the level of the iliac crest to the 4th lumbar vertebra and the quadratus lumborum muscle was visualized on the transverse process of the 4th lumbar vertebra at the point where the anterior abdominal wall muscles end. The needle was advanced in-plane between the quadratus lumborum muscle and the erector spinae-latissimus dorsi muscles (QLB2) located on the posterior-superior side of this muscle, and 0.15 ml/kg 0.25% bupivacaine was injected under the thoracolumbar fascia located between these two muscles. Then, the needle was advanced towards the quadratus lumborum and the psoas major (QLB3) muscle located on the anterior-inferior side, and 0.15 ml/kg 0.25% bupivacaine was injected between these two muscles.This procedure was applied to the patient bilaterally.
  Interventions: Procedure: Quadratus Lumborum Block (QLB); Drug: quadratus lumborum block using bupivacaine
- Transversus Abdominis Plane Group (TAPB) (Active Comparator): Transversus abdominis plane block was performed with the patient lying in the supine position via an oblique subcostal approach from the anterior abdominal wall. After skin asepsis of the anterior abdominal wall was provided with 10% polyvinylpyrrolidone-iodine, the linear ultrasound probe was placed parallel to the subcostal border at the level of the xiphoid bone and the subcutaneous fat tissue, rectus abdominis muscle and transversus abdominis muscle were visualized, respectively. A 10 cm 20G needle (BRAUN Stimuplex Ultra 360, GERMANY) was advanced towards the transversus abdominis muscle fascia with the in-plane technique and 0.3 ml/kg 0.25% bupivacaine was injected into this area.This procedure was performed bilaterally.
  Interventions: Procedure: transversus abdominis plane block; Drug: transversus abdominis plane block using bupivacaine

INTERVENTIONS:
Procedure: transversus abdominis plane block — Transversus abdominis plane block was performed with the patient lying in the supine position via an oblique subcostal approach from the anterior abdominal wall. After skin asepsis of the anterior abdominal wall was provided with 10% polyvinylpyrrolidone-iodine, the linear ultrasound probe was placed parallel to the subcostal border at the level of the xiphoid bone and the subcutaneous fat tissue, rectus abdominis muscle and transversus abdominis muscle were visualized, respectively. A 10 cm 20G needle (BRAUN Stimuplex Ultra 360, GERMANY) was advanced towards the transversus abdominis muscle fascia with the in-plane technique and 0.3 ml/kg 0.25% bupivacaine was injected into this area.This procedure was performed bilaterally.
  Arms: Transversus Abdominis Plane Group (TAPB)
Procedure: Quadratus Lumborum Block (QLB) — Quadratus lumborum block; after the patient was lying in the lateral decubitus position and skin asepsis of the posterior abdominal wall was provided with 10% polyvinylpyrrolidone-iodine, the ultrasound probe was moved from the level of the iliac crest to the 4th lumbar vertebra and the quadratus lumborum muscle was visualized on the transverse process of the 4th lumbar vertebra at the point where the anterior abdominal wall muscles end. The needle was advanced in-plane between the quadratus lumborum muscle and the erector spinae-latissimus dorsi muscles (QLB2) located on the posterior-superior side of this muscle, and 0.15 ml/kg 0.25% bupivacaine was injected under the thoracolumbar fascia located between these two muscles. Then, the needle was advanced towards the quadratus lumborum and the psoas major (QLB3) muscle located on the anterior-inferior side, and 0.15 ml/kg 0.25% bupivacaine was injected between these two muscles.This procedure was applied to the patient bilaterally.
  Arms: Quadratus Lumborum Group (QLB)
Drug: quadratus lumborum block using bupivacaine — The needle was advanced in-plane between the quadratus lumborum muscle and the erector spinae-latissimus dorsi muscles (QLB2) located on the posterior-superior side of this muscle, and 0.15 ml/kg 0.25% bupivacaine was injected under the thoracolumbar fascia located between these two muscles. Then, the needle was advanced towards the quadratus lumborum and the psoas major (QLB3) muscle located on the anterior-inferior side, and 0.15 ml/kg 0.25% bupivacaine was injected between these two muscles.This procedure was applied to the patient bilaterally.
  Arms: Quadratus Lumborum Group (QLB)
Drug: transversus abdominis plane block using bupivacaine — A 10 cm 20G needle (BRAUN Stimuplex Ultra 360, GERMANY) was advanced towards the transversus abdominis muscle fascia with the in-plane technique and 0.3 ml/kg 0.25% bupivacaine was injected into this area.This procedure was performed bilaterally.
  Arms: Transversus Abdominis Plane Group (TAPB)

SUMMARY:
Midline incisions provide easy, rapid and excellent exposure of the abdominal cavity and are particularly used for complex, diagnostic or emergency procedures.

However, midline incisions transect the nerve fibers passing in the mediocaudal direction of the abdominal wall, which causes more postoperative pain than other incisions.

Postoperative pain and delayed return of bowel function are thought to be the main factors that prevent early recovery and discharge.

or surgical procedures where parietal pain is the main component of postoperative pain, TAPB can be used as a simple and effective analgesic technique with the added advantage of preserved motor and bladder function.

Quadratus lumborum block can be used as an analgesic technique in all surgeries such as proctosigmoidectomy, hip surgery, above-knee amputation, abdominal hernia repair, breast reconstruction, colostomy closure, radical nephrectomy, lower extremity vascular surgery, total hip arthroplasty, laparotomy and colectomy.

Our study aimed to compare the effects of bilateral oblique subcostal TAPB with bilateral QLB2 and QLB3 performed under ultrasound guidance in midline incision laparotomies on total opioid requirement in the first 24 hours postoperatively, early postoperative pain intensity, time to first rescue analgesic requirement, nausea, vomiting and pruritus.

To evaluate this hypothesis, we compared TAPB and QLB in a prospective, randomized, single-center clinical study. The primary endpoint of our study was the comparison of total morphine consumption in the first 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Laparotomy with midline incision
* General anesthesia will be applied
* 18-70 years old
* ASA 1-3
* BMI of 18-30 kg/m2
* Literate
* Without cognitive impairment
* Patients who approved the informed consent form

Exclusion Criteria:

* Under 18 years old
* Over 70 years old
* ASA 4 and above
* Cognitive impairment
* İlliteracy
* Vision and hearing problem
* Infection at the injection site
* Coagulopathy
* Peripheral neuropathy
* Local anesthetic allergy
* Patients who do not want to be included in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Our study aimed to compare the effects of bilateral oblique subcostal TAPB with bilateral QLB2 and QLB3 performed under ultrasound guidance in midline incision laparotomies on total opioid requirement in the first 24 hours postoperatively | Within 24 hours after surgery
  All patients were extubated after the block was performed. All patients were given 1 mg bolus 10 min lock time IV morphine (Morphine Hydrochloride, OSEL Drug) connected to the PCA device (BodyGuard 575i Pain Manager, TARMED). If the morphine given with the PCA device was not sufficient as an analgesic, patients were given 1 gr IV paracetamol infusion (the dose was adjusted so that the paracetamol dose did not exceed a maximum of 4 grams per day). If the VAS was still >4 at 1 hour after paracetamol, the patient was administered 50 mg IV dexketoprofen (NSAID) (the dexketoprofen dose was adjusted to a maximum of 150 milligrams per day).he amount of opioids used and requested by the patients was recorded as the amount of PCA medication at the 15th minute, 2nd, 4th, 8th, 12th, 16th and 24th hours, as how much opioids they requested or used at the specified time intervals. For example, the amount of opioid used between the 15th minute and the 2nd hour was recorded at the 2nd hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Background] Mrunalini P, Raju NV, Nath VN, Saheb SM. Efficacy of transversus abdominis plane block in patients undergoing emergency laparotomies. Anesth Essays Res. 2014 Sep-Dec;8(3):377-82. doi: 10.4103/0259-1162.143153. PMID 25886339
- [Background] Liang SS, Ying AJ, Affan ET, Kakala BF, Strippoli GF, Bullingham A, Currow H, Dunn DW, Yeh ZY. Continuous local anaesthetic wound infusion for postoperative pain after midline laparotomy for colorectal resection in adults. Cochrane Database Syst Rev. 2019 Oct 19;10(10):CD012310. doi: 10.1002/14651858.CD012310.pub2. PMID 31627242
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=quadratus+lumborum+block